CLINICAL TRIAL: NCT06090890
Title: Safety and Efficacy of Low Dose Colchicine or Prednisone Combining With Standard Drug in Patients With Recurrent In-stent Restenosis: a Prospective, Randomized, Open-label Trial
Brief Title: Anti-inflammatory Therapy for Recurrent In-stent Restenosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Principal Investigator, Qian Haiyan, Director，Clinical Professor, Fu Wai Hospital, Beijing, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-GSP-GG-32
Record Dates: First submitted 2023-10-15; First posted 2023-10-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-09

CONDITIONS: In-stent Restenosis
Keywords: Anti-inflammatory therapy; In-stent Restenosis; Colchicine; Prednisone
MeSH Terms: interventions — Colchicine; Prednisone; Aspirin; Purinergic P2Y Receptor Antagonists; Hypolipidemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Active Comparator): DAPT (aspirin+1 P2Y12 receptor antagonist) + Lipid-lowering drugs + hypoglycemic drugs and hypotensive drugs (if necessary)
  Interventions: Drug: Aspirin; Drug: P2Y12 Receptor Antagonist; Drug: Lipid-lowering drug
- Colchicine group (Experimental): DAPT (aspirin+1 P2Y12 receptor antagonist) + Lipid-lowering drugs + hypoglycemic drugs and hypotensive drugs (if necessary) + Colchicine (0.5mg QD, orally)
  Interventions: Drug: Colchicine; Drug: Aspirin; Drug: P2Y12 Receptor Antagonist; Drug: Lipid-lowering drug
- Prednisone group (Experimental): DAPT (aspirin+1 P2Y12 receptor antagonist) + Lipid-lowering drugs + hypoglycemic drugs and hypotensive drugs (if necessary) + Prednisone (0.5mg/kg QD, orally)
  Interventions: Drug: Prednisone; Drug: Aspirin; Drug: P2Y12 Receptor Antagonist; Drug: Lipid-lowering drug

INTERVENTIONS:
Drug: Colchicine — Add 0.5mg QD orally and start using it within 48 hours after intervention.
  Arms: Colchicine group
Drug: Prednisone — 0.5mg/kg QD orally and the dosage was reduced at a rate of 5mg/d per month until 5-10mg/d, maintained for 1 year after PCI.
  Arms: Prednisone group
Drug: Aspirin — Patients who have re-implanted DES should receive aspirin for at least 1 year after intervention; Patients who have underwent DEB expansion should apply aspirin for at least 3 months after intervention.
  Other Names: Acetylsalicylic Acid
Drug: P2Y12 Receptor Antagonist — Patients who have re-implanted DES should receive 1 P2Y12 receptor antagonist for at least 1 year after intervention; Patients who have underwent DEB expansion should apply the P2Y12 receptor antagonist for at least 3 months after intervention.
Drug: Lipid-lowering drug — Formulate the lipid-lowering drug regimen with LDL-C<1.4mmol/L as the target on the basis of moderate intensity or above statins.

SUMMARY:
This study is aimed at making a comparison of the safety and efficacy of standard drug therapy (control group), standard drugs combined with lose-dose colchicine therapy (colchicine group) and standard drug combined with prednisone therapy (prednisone group) in patients with coronary heart disease who suffered from recurrent In-stent restenosis (RISR).

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, blinded-endpoint evaluation, single-center Study. A total of 252 RISR patients are planned to be enrolled in Fuwai Hospital, China. Then those included subjects will be randomized to standard drug therapy (control group), standard drugs combined with lose-dose colchicine therapy (colchicine group) and standard drug combined with prednisone therapy (prednisone group). The primary endpoint of the current study is target lesion ISR confirmed by coronary angiography for 12 months, and the secondary endpoint is Major adverse cardiovascular events (MACE: a composite of death, non-fatal myocardial infarction, non-fatal stroke, and target vascular revascularization) and each MACE component, target lesion revascularization, or other coronary artery disease revascularization for 12 months. The safety endpoint is adverse reactions to colchicine, adverse reactions of prednisone, or discontinued medication due to adverse reactions. In summary, the present study is to provide new evidence and strategy about anti-inflammatory therapy for recurrent In-stent restenosis after coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

1. CAD patients over 18 years old;
2. At least one coronary artery lesion meets the RISR criteria: target lesion ≥ 2 ISRs (stenosis of lumen diameter within the stent segment and within 5mm near and far of the stent ≥ 50%);
3. Intended intervention treatment for RISR lesions;
4. Acceptable for standard secondary prevention drug therapy for coronary heart disease, including dual antiplatelet therapy (DAPT) and statins;
5. Willing to participate in the trial and complete follow-up, signing an informed consent form approved by the ethics committee

Exclusion Criteria:

1. The previous interventional treatment situation is unknown;
2. The mechanism of intracavitary imaging to clarify ISR is operator-related (poor stent adhesion, incomplete dilation, and stent fracture);
3. Clearly diagnose vascular inflammatory diseases or connective tissue diseases (including arteritis, Behcet's disease, systemic lupus erythematosus, etc.) involving the coronary artery;
4. Immunosuppressive drugs, including glucocorticoids, have been used in the past 30 days;
5. There are contraindications to the use of prednisone or colchicine, including: serious infectious diseases, including active infection, hepatitis B, hepatitis C or AIDS patients; Hematological diseases, such as thrombocytopenia, severe anemia, leukemia, etc; Uncontrolled diabetes; Severe liver and kidney function damage; Active peptic ulcer or gastrointestinal bleeding; Severe osteoporosis (with previous pathological fractures); Inflammatory bowel disease or chronic diarrhea;
6. A history of malignant tumors within 3 years;
7. Cognitive impairment;
8. Not willing to participate or follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
target lesion ISR | 12 months after randomization
  target lesion ISR confirmed by coronary angiography for 12 months

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events | 12 months after randomization
  a composite of mortality, non-fatal myocardial infarction, non-fatal stroke and target vascular revascularization
target lesion revascularization | 12 months after randomization
  incidence of revascularization due to target lesion
other coronary artery disease revascularization | 12 months after randomization
  incidence of revascularization due to other coronary artery disease

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Qian, Principal Investigator — Fuwai Hospital, Beijing, China
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be securely stored and will be available only upon reasonable request and with approval from the study investigators, in accordance with BMJ Open's data-sharing policy.
Supporting Information: Study Protocol, SAP
Access Criteria: De-identified individual participant data will be available only upon reasonable request and with approval from the study investigators, in accordance with BMJ Open's data-sharing policy.

REFERENCES:
- [Derived] Yu M, Jiang Y, Song Z, Wei ZY, Tan F, Liu X, Zhang X, Zhu F, Shi Y, Huang J, Yang WX, Qian HY. Anti-inflammatory therapy for recurrent in-stent restenosis (AI-ISR): study protocol for a prospective, randomised, open-label, multicentre clinical trial. BMJ Open. 2025 Oct 27;15(10):e092235. doi: 10.1136/bmjopen-2024-092235. PMID 41145262